CLINICAL TRIAL: NCT00354510
Title: Randomised, Double-blind, Placebo-controlled Study of Topical GW842470X Formulation in Adults With Moderate Atopic Dermatitis
Brief Title: Topical GW842470X In Adults Patients With Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TPD103280
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-03

CONDITIONS: Atopic Dermatitis; Dermatitis, Atopic
Keywords: atopic dermatitis; GW842470X; PDE4 inhibitor
MeSH Terms: conditions — Dermatitis, Atopic

INTERVENTIONS:
Drug: GW842470X cream

SUMMARY:
The purpose of this study is to investigate the clinical efficacy of 3% (w/w) GW842470X cream applied to involved skin of adult patients with moderate atopic dermatitis using the Eczema Area Severity Index (EASI) assessment of disease severity and to investigate the safety of and tolerability of 3% GW842470X cream on diseased skin of adult patients.

ELIGIBILITY:
Inclusion criteria:

* Moderate atopic dermatitis patients (IGA=3).
* The disease involvement must be >5% of body surface area.
* Female patients of child-bearing potential must use an appropriate method of contraception.

Exclusion criteria:

* Patients with any active skin disease other than atopic dermatitis will not be eligible.
* Patients who have had systemic treatment for atopic dermatitis or other topical or transdermal treatments (such as nicotine, hormone replacement therapies) within 14 days prior to first application of study medication and/or topical treatment with tar, any corticosteroid, topical immunomodulators or oral treatment with any corticosteroids within 10 days prior to first application and/or oral anti-histamines within 5 days of the first dose.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190
Dates: Start 2006-03

PRIMARY OUTCOMES:
Clinical efficacy of 3% GW842470X cream applied to involved skin of adult patients with moderate atopic dermatitis using the Eczema Area Severity Index (EASI).

SECONDARY OUTCOMES:
Safety and tolerability of 3% GW842470X cream
Clinical efficacy using SCORing Atopic Dermatitis score & Investigators Global Assessment Scale
Symptoms: pruritus & sleep loss
Characterize systemic exposure to GW842470X following 21 days treatment.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- Germany (7):
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Mahlow, Brandenburg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Duelmen, Lower Saxony
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Schenefeld, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
- Netherlands (3):
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Utrecht